CLINICAL TRIAL: NCT01004809
Title: An Open Label, Multi-centre, Non-interventional Post-marketing Surveillance to Monitor the Safety and Effectiveness of AVODART® Administered in Korean Androgenetic Alopecia Patients According to the Prescribing Information
Brief Title: AVODART® Alopecia Post-marketing Surveillance (PMS)
Acronym: AVODART®PMS
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113797
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Alopecia
Keywords: Dutasteride
MeSH Terms: conditions — Alopecia | interventions — Dutasteride

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dutasteride: Patients administrated dutasteride with male hair loss
  Interventions: Drug: Dutasteride

INTERVENTIONS:
Drug: Dutasteride — Basically there is no treatment allocation. Subjects who would be administered of dutasteride at their physicians' discretion will be enrolled. Dosage regimen will be recommended according to the prescribing information. Subjects will be enrolled consecutively.

SUMMARY:
Post-marketing surveillance(PMS) to monitor the safety and effectiveness of dutasteride in Korean androgenetic alopecia patients

DETAILED DESCRIPTION:
An open label, multi-centre, non-interventional post-marketing surveillance to monitor the safety and effectiveness of dutasteride administered in Korean androgenetic alopecia patients according to the prescribing information

ELIGIBILITY:
Inclusion Criteria:

* Men (18-41 years of age) with male pattern hair loss (androgenetic alopecia)
* Subjects with no experience of treatment using dutasteride
* Subjects who the investigator believes that they can and will comply with the requirements of the protocol
* Subjects who prescribed with dutasteride according to the Prescribing Information

Exclusion Criteria:

* Considering the nature of observational study, GSK Korea encourages the doctors participating in this study to enrol the subjects prescribed with dutasteride following the locally approved Prescribing Information. Subject who give informed consent is enrolled. However, if institution waives the requirement for informed consent, informed consent is not required. In this case, monitoring does not proceed.

Ages: 18 Years to 41 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients administrated dutasteride with male pattern hair loss (androgenetic alopecia)
Sampling Method: Probability Sample
Enrollment: 712 (Actual)
Dates: Start 2010-04-29; Primary Completion 2012-12-01 (Actual); Study Completion 2012-12-21 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse event after dutasteride administration | 2 years

SECONDARY OUTCOMES:
Occurrence of unexpected adverse drug reaction after dutasteride administration | 2 years
Occurrence of serious adverse events after dutasteride administration | 2 years
Effectiveness of dutasteride judged by a physician | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Daejeon, South Korea